CLINICAL TRIAL: NCT00274833
Title: A Phase II Trial of Erlotinib With Temozolomide and Concurrent Radiation Therapy Post-Operatively in Patients With Newly Diagnosed Glioblastoma Multiforme
Brief Title: Radiation Therapy, Temozolomide, and Erlotinib in Treating Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: David Peereboom (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, David Peereboom, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE3304; P30CA043703 (NIH); CASE3304 (Other: Case Comprehensive Cancer Center); CCF-6320 (Other: Cleveland Clinic IRB)
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: CNS Tumor, Adult
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Erlotinib Hydrochloride; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiation Therapy, Temozolomide, and Erlotinib (Experimental)
  Interventions: Drug: erlotinib hydrochloride; Drug: temozolomide; Radiation: radiation therapy

INTERVENTIONS:
Drug: erlotinib hydrochloride — Erlotinib is available as 25 mg, 100 mg, and 150 mg tablets. It should be administered orally once daily at the prescribed dose specified in the clinical study protocol per dose escalation schema. Preferably, erlotinib should be taken in the morning with up to 200 mL of water at least 1 hour before or 2 hours after a meal.
  Other Names: Tarceva
Drug: temozolomide — TMZ is supplied in white opaque, preservative-free, two piece hard gelatin capsules of the following sizes: 100mg capsules, 20mg capsules, and 5mg capsules. TMZ will be a once a day orally administered (75 mg/m2 x BSA x 42 days)set of capsules taken at least two hours after and one hour before a meal.
  Other Names: Temodar
Radiation: radiation therapy — Concomitant focal RT will be delivered once daily at 2 Gy per fraction, 5 d/wk, for a total of 60 Gy. (6 weeks) as mentioned in therapeutic modalities.
  Other Names: RT

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving radiation therapy together with temozolomide and erlotinib after surgery may kill any remaining tumor cells.

PURPOSE: This phase II trial is studying how well giving radiation therapy together with temozolomide and erlotinib works in treating patients with newly diagnosed glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the progression-free survival and overall survival of patients with newly diagnosed glioblastoma multiforme treated with adjuvant radiotherapy, temozolomide, and erlotinib hydrochloride.
* Evaluate the toxicity of this regimen in these patients.

OUTLINE: This is a non-randomized study.

Patients receive oral temozolomide once daily on days 1-42 and undergo concurrent radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-40. Four weeks after completion of radiotherapy and temozolomide, patients receive oral temozolomide once daily on days 1-5. Treatment with temozolomide repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity. Patients also receive oral erlotinib hydrochloride once daily beginning on day 1 of radiotherapy and continuing in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven glioblastoma multiforme

  * Newly diagnosed disease
* Has undergone diagnostic biopsy or surgical resection within the past 28 days

PATIENT CHARACTERISTICS:

* ECOG 0-2
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin > 9 g/L
* Serum creatinine and total serum bilirubin < 1.5 times upper limit of normal (ULN)
* AST or ALT < 2.5 times ULN
* Alkaline phosphatase < 2.5 times ULN
* No other severe underlying disease (including HIV or chronic hepatitis B or C infection)
* Fertile patients must use effective contraception
* Not pregnant or nursing
* No medical condition that could interfere with the oral administration of temozolomide or erlotinib hydrochloride
* No other malignancy within the past 3 years with the exception of surgically cured carcinoma in situ of the cervix, nonmelanoma skin cancer, or adequately treated stage I or II cancer from which the patient is in complete remission
* No active infection
* No other condition that would preclude ability of the patient to be followed closely at the Cleveland Clinic

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy or chemotherapy for this cancer
* No prior cranial radiotherapy
* No concurrent enzyme-inducing anti-epileptic drugs
* No prior temozolomide or erlotinib hydrochloride
* No other concurrent antineoplastic therapy
* No concurrent filgrastim (G-CSF) or sargramostim (GM-CSF) during chemotherapy
* No concurrent electron, particle, or implant boost radiotherapy
* No concurrent radiosurgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2005-10; Primary Completion 2007-10 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | at 6 months

SECONDARY OUTCOMES:
Progression Free Survival | at 1 yr
Number of patients that experience toxicity (CTCAE V2) | at 6 months
Overall Survival | date of final follow up visit

CONTACTS AND LOCATIONS:
Overall Officials: David M. Peereboom, MD, Study Chair — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States